CLINICAL TRIAL: NCT05824039
Title: Safety and Efficacy of the Short Daily Administration of Nitraria Retusa Extract in Overweight and Obese Participants. .
Brief Title: Safety and Efficacy of Medicinal Plant Extract in Overweight and Obese Participants.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laouani Aicha (Other)
Collaborators: Faculty of Medicine, Sousse (Other); Centre Hôpital Universitaire Farhat Hached (Other); Université de Sousse (Other); University of Tsukuba (Other)
Responsible Party: Sponsor-Investigator, Laouani Aicha, Assistant Professor PHD, Head of the common Services unit for Research , biophysics Laboratory, Faculty of Medicine, Sousse
Organization: Faculty of Medicine, Sousse (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEFMS 34/2019
Record Dates: First submitted 2023-04-11; First posted 2023-04-21 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Overweight; Obesity
Keywords: Medicinal plants; Anti-lipidimic agents; Infusion
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental 1: low dose group (Experimental): Tea infusion which contain 5 mg of flavonoids, (low dose of flavonoids treatment quantification) oral administration , once daily.
  Interventions: Dietary Supplement: Tea infusion
- Experimental 2 : high dose group (Experimental): Tea infusion which contain 20 mg of flavonoids, ( high dose of flavonoids Treatment quantification) oral administration , once daily .
  Interventions: Dietary Supplement: Tea infusion

INTERVENTIONS:
Dietary Supplement: Tea infusion — Tea infusion: The aerial parts of the medicinal plant were dried, then, they were powdered in a rotating knife grinder. The herbs were taken as tea infusion by the oral route. The powder was added to 100 ml of boiling water and the tea infusion was taken once time a day at the bed time and it was repeated for 10 days.

SUMMARY:
The purpose of this randomized , double -blind clinical trial is to evaluate the efficacy and safety of a daily administration of Nitraria retusa extract in overweight and obese participants, during 10 days.

DETAILED DESCRIPTION:
Medicinal plants are widely used for their accessibility, safety and effectiveness and may be an excellent alternative strategy for developing future drugs with minor adverse effects. Several studies concerning the potential of bioactive components in plants and food products and their link to many diseases including, diabetes, cardiovascular disease and obesity.

Nitraria retusa is a salt-tolerant plant that belongs to the Nitrariaceae family. It is particularly distributed in Asia, China, North Africa, Russia and Europe.It grows in the southern part of Tunisia and it is locally known as Ghardaq. The leaves serve as supplement for the tea and are used as poultice. Fresh leaves of Nitraria retusa have been used in traditional medicine in case of poisoning, upset stomach, ulcers, gastritis, enteritis, heartburn, colitis, and colonic abdominal pain.

Moreover, anticancer, antioxidant, antiviral and antimicrobial activities of N. retusa have been reported .Several reports evinced that the leaf of Nitraria retusa contains high amounts of tannins, alkaloids, steroids and flavonoids, which could be responsible for its beneficial effects . Previous studies have demonstrated the effect of Nitraria retusa extract in obese mice against high fat diet through lowering glucose and triglycerides and the enhancement of the lipid metabolism in liver.

The purpose of this study was to evaluate the efficacy and safety of short daily administration of Nitraria retusa extract in lipid profile in overweight and obese patients, during 10 days.

This study will be carried out in 2 departments: the laboratory of biophysics of the Faculty of Medicine of Sousse and Endocrinology and diabetology of CHU Farhat Hached Sousse ,Tunisia. At day 0 and day 10 all the population will benifit of biological assessment which include:

* Biochimical parameters

  * Complete lipid profile (Total Cholesterol (T-C), High-density Lipoprotein (HDL) Low-density Lipoprotein (LDL) and Triglycerides( TG) .
  * Blood sugar
  * Liver Function Test : Alkaline phosphatase (ALP), gamma-glutamyltransferase (G-GT), albumin, Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), total ( TB) and direct bilirubin (DB).
  * Renal Function Test : Serum Creatinine, urea
  * Inflammatory assessment: Reactive protein C
* Hematological parameters : (Red blood cells (RBC), White blood cell (WBC), Platelet, Hemoglobin and Hematocrit).

All Population will be randomized :Participant will be assigned to one of two treatments (low dose flavonoids or high dose flavonoids ). The diatry supplement :Nitraria retusa infusion will be prescribed at a quantity of powder which contained 5 mg of flavonoids or which contained 20 mg of flavonoids , added to 100 ml of boiling water and will be taken once a day at a bed time for 10 consecutive days.

Statistical analysis Data entry and analysis will be performed using SPSS 22.0 for Windows(IBM Corp., NY, USA ). Results will be considered significant at p < 0.05 Normal distributions of the data will be assessed by Shapiro-Wilk test. Within-group differences in the biological parameters before and after the intervention will be compared using paired t-test when data are normally distributed and Wilcoxon Signed Rank Test when data are not normaly distrubuted. Between-group differences (low dose vs high dose) in the parameters will be assessed by independent samples t-test (parametric and equal variances), Welch's t-test (unequal variances) and Mann-Whitney U test (nonparametric)

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* age range of 18 and 75 years
* BMI >25 kg/ m^2

Exclusion Criteria:

* Hypertension
* Diabetes
* Asthma
* Smoking
* Professional athletic
* Pregnancy and breast feeding
* Participant with medical or psychiatric disorder or chronic pathology,
* Participant with eating disorder, food allergies.
* Participant with a history of cardiovascular disease,
* Participant with medication known to affect lipid metabolism,
* Participant with major gastrointestinal problems.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2021-03-20 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2022-04-08 (Actual)

PRIMARY OUTCOMES:
Change in serum Triglycerides (TG) levels | 10 days
  To evaluate the efficacy of 20 mg of flavonoids in reducing serum TG compared with low dose group ( 5 mg of flavonoids) after 10 days administration .
Change in serum High Density Lipoprotein Cholesterol (HDL-C) levels | 10 days
  To evaluate the efficacy of 20 mg of flavonoids in increasing HDL-C levels compared with low dose group ( 5 mg of flavonoids) after 10 days administration
Change in Total Cholesterol ( TC) levels | 10 days
  To evaluate the efficacy of 20 mg of flavonoids in reducing TC levels compared with low dose group ( 5 mg of flavonoids) after 10 days administration.
Change in Low Density Lipoprotein Cholesterol (LDL-C) levels | 10 days
  To evaluate the efficacy of 20 mg of flavonoids in reducing LDL-C levels compared with low dose group ( 5 mg of flavonoids) after 10 days administration

SECONDARY OUTCOMES:
no change from baseline in Alkaline phosphatase levels | 10 days
no change from baseline in Aspartate aminotransferase levels. | 10 days
no change from baseline in Alanine aminotransferase levels. | 10 days
no change from baseline in gamma-glutamyltransferase levels. | 10 days
no change from baseline in Albumin levels . | 10 days
no change from baseline in total bilirubin levels | 10 days
no change from baseline in direct bilirubin levels | 10 days
no change from baseline in urea levels | 10 days
no change from baseline in creatinine levels | 10 days
no change from baseline in fasting blood glucose levels | 10 days
no change from baseline in Red blood cells levels | 10 days
no change from baseline in White blood cells levels | 10 days
no change from baseline in Hemoglobin levels | 10 days
no change from baseline in Hematocrit levels | 10 days
no change from baseline in Platelets levels | 10 days
no change from baseline in Hemodynamic indicators: heart rate and blood pressure : systolic blood pressure and diastolic blood pressure | 10 days
Adverse events | 10 days
  Adverse events reported

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine of Sousse, 4000 Tunisia, Sousse, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boubaker J, Bhouri W, Ben Sghaier M, Ghedira K, Dijoux Franca MG, Chekir-Ghedira L. Ethyl acetate extract and its major constituent, isorhamnetin 3-O-rutinoside, from Nitraria retusa leaves, promote apoptosis of human myelogenous erythroleukaemia cells. Cell Prolif. 2011 Oct;44(5):453-61. doi: 10.1111/j.1365-2184.2011.00772.x. PMID 21951288
- [Background] Boubaker J, Bhouri W, Sghaier MB, Bouhlel I, Skandrani I, Ghedira K, Chekir-Ghedira L. Leaf extracts from Nitraria retusa promote cell population growth of human cancer cells by inducing apoptosis. Cancer Cell Int. 2011 Oct 31;11(1):37. doi: 10.1186/1475-2867-11-37. PMID 22040460
- [Background] Chaabane M, Koubaa M, Soudani N, Elwej A, Grati M, Jamoussi K, Boudawara T, Ellouze Chaabouni S, Zeghal N. Nitraria retusa fruit prevents penconazole-induced kidney injury in adult rats through modulation of oxidative stress and histopathological changes. Pharm Biol. 2017 Dec;55(1):1061-1073. doi: 10.1080/13880209.2016.1278455. PMID 28198206
- [Background] Hashempur MH, Mosavat SH, Heydari M, Shams M. Medicinal plants' use among patients with dyslipidemia: an Iranian cross-sectional survey. J Complement Integr Med. 2018 Nov 3;16(3):/j/jcim.2019.16.issue-3/jcim-2018-0101/jcim-2018-0101.xml. doi: 10.1515/jcim-2018-0101. PMID 30391934
- [Background] Zar Kalai F, Han J, Ksouri R, Abdelly C, Isoda H. Oral administration of Nitraria retusa ethanolic extract enhances hepatic lipid metabolism in db/db mice model 'BKS.Cg-Dock7(m)+/+ Lepr(db/)J' through the modulation of lipogenesis-lipolysis balance. Food Chem Toxicol. 2014 Oct;72:247-56. doi: 10.1016/j.fct.2014.07.029. Epub 2014 Jul 30. PMID 25086370
- [Background] Rjeibi I, Feriani A, Hentati F, Hfaiedh N, Michaud P, Pierre G. Structural characterization of water-soluble polysaccharides from Nitraria retusa fruits and their antioxidant and hypolipidemic activities. Int J Biol Macromol. 2019 May 15;129:422-432. doi: 10.1016/j.ijbiomac.2019.02.049. Epub 2019 Feb 8. PMID 30742925
- [Background] Zar Kalai F, Han J, Ksouri R, El Omri A, Abdelly C, Isoda H. Antiobesity Effects of an Edible Halophyte Nitraria retusa Forssk in 3T3-L1 Preadipocyte Differentiation and in C57B6J/L Mice Fed a High Fat Diet-Induced Obesity. Evid Based Complement Alternat Med. 2013;2013:368658. doi: 10.1155/2013/368658. Epub 2013 Dec 3. PMID 24367387